CLINICAL TRIAL: NCT02790580
Title: Dose-dense Doxorubicin/Cyclophosphamide With Intermittent Low-dose Sunitinib as Neoadjuvant or First-line Palliative Treatment of Newly Diagnosed HER2 Negative Breast Cancer Patients With Measurable Primary Breast Tumor
Brief Title: Dose-dense Doxorubicin/Cyclophosphamide With Intermittent Low-dose Sunitinib in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR01/01/16; 2016/00327 (Other: NHG DSRB)
Record Dates: First submitted 2016-05-30; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-dense doxorubicin/cyclophosphamide (Active Comparator): Doxorubicin 60mg/m2 day 1, every 2 weeks x 4 cycles, Cyclophosphamide 600mg/m2 day1, every 2 weeks x 4 cycles, Subcutaneous pegfilgrastim 6mg, 24-36 hours after doxorubicin/cyclophosphamide
  Interventions: Drug: Dose-dense doxorubicin/cyclophosphamide
- Dose-dense doxorubicin/cyclophosphamide + sunitinib (Experimental): Doxorubicin 60mg/m2 day 1, every 2 weeks x 4 cycles, Cyclophosphamide 600mg/m2 day1, every 2 weeks x 4 cycles, Subcutaneous pegfilgrastim 6mg, 24-36 hours after each cycle of doxorubicin/cyclophosphamide, Oral sunitinib 12.5mg daily for 7 days prior to cycle 1 ddAC (days -7 to 0), Oral sunitinib 12.5mg daily for 5 days prior to cycle 2, 3, 4 ddAC (days 10-14 of preceding cycle)
  Interventions: Drug: Dose-dense doxorubicin/cyclophosphamide + sunitinib

INTERVENTIONS:
Drug: Dose-dense doxorubicin/cyclophosphamide + sunitinib — Doxorubicin 60mg/m2 day 1, every 2 weeks x 4 cycles Cyclophosphamide 600mg/m2 day1, every 2 weeks x 4 cycles Subcutaneous pegfilgrastim 6mg, 24-36 hours after each cycle of doxorubicin/cyclophosphamide Oral sunitinib 12.5mg daily for 7 days prior to cycle 1 ddAC (days -7 to 0) Oral sunitinib 12.5mg daily for 5 days prior to cycle 2, 3, 4 ddAC (days 10-14 of preceding cycle)
  Lumpectomy or mastectomy with sentinel lymph node biopsy or axillary lymph node clearance as appropriate should be considered after completing four cycles of chemotherapy for curative intent in non-metastatic patients and for local control for patients with metastatic disease.
  Arms: Dose-dense doxorubicin/cyclophosphamide + sunitinib
Drug: Dose-dense doxorubicin/cyclophosphamide — Doxorubicin 60mg/m2 day 1, every 2 weeks x 4 cycles Cyclophosphamide 600mg/m2 day1, every 2 weeks x 4 cycles Subcutaneous pegfilgrastim 6mg, 24-36 hours after each cycle of doxorubicin/cyclophosphamide
  Lumpectomy or mastectomy with sentinel lymph node biopsy or axillary lymph node clearance as appropriate should be considered after completing four cycles of chemotherapy for curative intent in non-metastatic patients and for local control for patients with metastatic disease.
  Arms: Dose-dense doxorubicin/cyclophosphamide

SUMMARY:
Background: The investigators previously studied the addition of low-dose, short-course sunitinib to pre-operative chemotherapy in the neoadjuvant setting in newly diagnosed breast cancer patients with measurable primary breast tumor in a phase Ib/II study at the National University Cancer Institute, Singapore. These data showed that the addition of sunitinib improved tumor vascularization as hypothesized with enhanced short-term treatment response. However, pathological complete response rate after 4 cycles of chemotherapy was not superior to standard chemotherapy, and may be attributed to dose delays from increased myelosuppression with the addition of sunitinib. The investigators hypothesize that this promising regimen may be further optimized with the use of growth factor support. The investigators thus plan to study the addition of low-dose, shortcourse sunitinib to dose-dense doxorubicin/cyclophosphamide (ddAC) administered every 14 days, supported by pegfilgrastim.

Aim: To confirm that the addition of 12.5mg sunitinib for 5-7 days can be added before each cycle of ddAC (delivered every 14 days, supported by pegfilgrastim) without compromising dose intensity, in phase II open label single arm part of the study, followed by a phase II randomized study to compare the pathological complete response rate of ddAC versus sunitinib + ddAC in stage I-III HER2 negative breast cancer patients in the neoadjuvant setting.

Methods:A single-centre study comprising two phases: a. Phase II open label single-arm study that will enroll newly diagnosed stage I-IV HER2 negative breast cancer patients receiving either neoadjuvant chemotherapy (stage I-III patients) or first-line palliative chemotherapy (stage IV patients). All patients will be treated with 4 cycles of ddAC at standard doses (60/600mg/m2) every 2 weeks, supported by subcutaneous pegfilgrastim 6mg, to be administered 24-36 hours after each dose of chemotherapy. Low dose sunitinib at 12.5mg daily orally will be administered for 7 days prior to cycle 1 ddAC, and for 5 days prior to each subsequent cycle of ddAC. b. Phase II randomized study that will enroll newly diagnosed stage I-III HER2 negative breast cancer patients receiving neoadjuvant chemotherapy before definitive breast cancer surgery. Eligible patients will be randomized 1:1 to 4 cycles of ddAC with or without intermittent sunitinib in patients with measurable primary breast cancer who are receiving preoperative chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is a major cause of morbidity and mortality both locally as well as globally. Approximately 10-15% of newly diagnosed breast cancer patients present with metastatic disease; in addition, a significant proportion of patients who initially present with non-metastatic disease relapse with distant metastases. These patients have no prospect for cure, and systemic therapy remains the mainstay of treatment. In the last few years, several targeted agents have been approved for the treatment of breast cancer. For example, the addition of bevacizumab, an anti-angiogenic agent, to chemotherapy has been shown to improve treatment outcome in metastatic HER2 negative breast cancer and possibly in the neoadjuvant treatment of triple negative breast cancers. Two classes of anti-angiogenic agents are currently available: monoclonal antibodies against vascular endothelial growth factor (VEGF), such as bevacizumab; and small molecule receptor tyrosine kinase inhibitors that target the intracellular tyrosine kinase domain of vascular endothelial growth factor receptor (VEGF-R), such as sunitinib and sorafenib.

Small molecule receptor tyrosine kinase inhibitors such as sunitinib and sorafenib are currently being evaluated in clinical trials. Although sunitinib and sorafenib are potent anti-angiogenic agents, the clinical data that has been reported thus far when combined with chemotherapy, has been less promising than what has been predicted in pre-clinical studies. One possible reason is that optimal scheduling of small molecule tyrosine kinase inhibitors with chemotherapy has not yet been determined. Preclinical observations have suggested that anti-angiogenic agents can 'normalize' tumor vasculature. Further continuous administration of anti-angiogenic agent ultimately results in destruction of tumor vasculature, starving the tumor and resulting in tumor necrosis. When combined with chemotherapy, this continuous scheduling may paradoxically result in reduced delivery of chemotherapy to the tumor, causing a relatively chemo-resistant state and may account for the less than optimal results from combination studies, which have largely employed the strategy of continuous dosing of the small molecule tyrosine kinase inhibitor. Intermittent dosing of a small molecule tyrosine kinase inhibitor prior to chemotherapy to transiently 'normalize' tumor vasculature, may make it more efficient for drug and oxygen delivery, and thus potentiate sensitivity to chemotherapy.

The investigators previously studied the addition of low-dose, short-course sunitinib to pre-operative chemotherapy in the neoadjuvant setting in newly diagnosed breast cancer patients with measurable primary breast tumor in a phase Ib/II study at the National University Cancer Institute, Singapore. The study data showed that the addition of sunitinib improved tumor vascularization as hypothesized with enhanced short-term treatment response. However, pathological complete response rate after 4 cycles of chemotherapy was not superior to standard chemotherapy, and may be attributed to dose delays from increased myelosuppression with the addition of sunitinib. The investigators hypothesize that this promising regimen may be further optimized with the use of growth factor support. The investigators thus plan to study the addition of low-dose, short-course sunitinib to dose-dense doxorubicin/cyclophosphamide administered every 14 days, supported by pegfilgrastim.

ELIGIBILITY:
Inclusion Criteria:

* Female, age ≥ 18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* T2-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with both diameters 2.0cm or greater as measured by caliper.
* Patients with synchronous breast tumors (ipsilateral or bilateral) may be enrolled, provided that none of the tumors is HER2 positive. Protocol-specific biopsy will be performed for each tumor, and each tumor will be assessed separately for pCR rate if the patient is non-metastatic
* Tumor must be HER2 negative by IHC (0 or 1+), or FISH (dual-probe HER2/CEP17 ratio <2.0 with average HER2 copy number <4.0 signals/cell)
* Patients must not have received prior chemotherapy or hormonal therapy for the treatment of breast cancer.
* ECOG performance 0 or 1.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  - Bone marrow: Absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L

  - Hepatic: Bilirubin ≤ 1.5 x upper limit of normal (ULN), ALT or AST ≤ 2.5x ULN, (or ≤5 X with liver metastases)

  - Renal: Creatinine ≤ 1.5x ULN
* Left ventricular ejection fraction ≥50%
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (e.g., intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Prior treatment for locally advanced or metastatic breast cancer.
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment, with exception of a synchronous HER2 negative breast cancer that is not metastatic
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Known history of systemic connective tissue diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis), vasculitidies (e.g., giant cell arteritis, Kawasaki disease, Wegener's granulomatosis, Churg-Strauss disease) or sickle cell disease.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | Post neoadjuvant chemotherapy (within 2-3 weeks after last dose of neoadjuvant chemotherapy)

SECONDARY OUTCOMES:
Pathological complete response rate | Post neoadjuvant chemotherapy (within 4-6 weeks after last dose of neoadjuvant chemotherapy)
Progression-free survival | 2 and 5 year post neoadjuvant chemotherapy/time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burstein HJ, Elias AD, Rugo HS, Cobleigh MA, Wolff AC, Eisenberg PD, Lehman M, Adams BJ, Bello CL, DePrimo SE, Baum CM, Miller KD. Phase II study of sunitinib malate, an oral multitargeted tyrosine kinase inhibitor, in patients with metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2008 Apr 10;26(11):1810-6. doi: 10.1200/JCO.2007.14.5375. Epub 2008 Mar 17. PMID 18347007
- [Background] Duda DG, Batchelor TT, Willett CG, Jain RK. VEGF-targeted cancer therapy strategies: current progress, hurdles and future prospects. Trends Mol Med. 2007 Jun;13(6):223-30. doi: 10.1016/j.molmed.2007.04.001. Epub 2007 Apr 25. PMID 17462954
- [Background] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Derived] Choo JRE, Jan YH, Ow SGW, Wong A, Lee MX, Ngoi N, Yadav K, Lim JSJ, Lim SE, Chan CW, Hartman M, Tang SW, Goh BC, Tan HL, Chong WQ, Yvonne ALE, Chan GHJ, Chen SJ, Tan KT, Lee SC. Serial Tumor Molecular Profiling of Newly Diagnosed HER2-Negative Breast Cancers During Chemotherapy in Combination with Angiogenesis Inhibitors. Target Oncol. 2022 May;17(3):355-368. doi: 10.1007/s11523-022-00886-x. Epub 2022 Jun 14. PMID 35699834
- [Derived] Yadav K, Lim J, Choo J, Ow SGW, Wong A, Lee M, Chan CW, Hartman M, Lim SE, Ngoi N, Tang SW, Ang Y, Chan G, Chong WQ, Tan HL, Tan SH, Goh BC, Lee SC. Immunohistochemistry study of tumor vascular normalization and anti-angiogenic effects of sunitinib versus bevacizumab prior to dose-dense doxorubicin/cyclophosphamide chemotherapy in HER2-negative breast cancer. Breast Cancer Res Treat. 2022 Feb;192(1):131-142. doi: 10.1007/s10549-021-06470-7. Epub 2021 Dec 20. PMID 34928481